CLINICAL TRIAL: NCT02983838
Title: Development of Biomarker With Neuroimaging : Research on Pathophysiology and Treatment in Depression Using Brain Derived Neurotrophic Factor (BDNF) and Amyloid Neuroimaging
Brief Title: Research on Pathophysiology and Treatment in Depression Using Brain Derived Neurotrophic Factor and Amyloid Neuroimaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Sungkyunkwan University (Other); Korea University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-12-009
Record Dates: First submitted 2016-04-13; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: Amyloid; BDNF; major depressive disorder; cognitive decline
MeSH Terms: conditions — Depressive Disorder, Major; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — blood specimen for pro-inflammatory cytokine and BDNF BDNF genotyping
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- depression with cognitive impairment: depression onset after 60 years old with subjective cognitive impairment
- depression without cognitive impairment: depression onset after 60 years old without subjective cognitive impairment
- normal control: older than 65 years, free from other neurocognitive disorder

SUMMARY:
Target of the research Based on change of Brain-derived neurotrophic factor and other pro-inflammatory cytokine along with symptom improvement following treatment, the investigators are trying to find the new treatment target molecule. The investigators will follow up the subjective and objective cognitive dysfunction with psychiatric symptom profiles and compare the neuroimaging related to these change.

DETAILED DESCRIPTION:
Recently the investigators reported the association between childhood trauma and refractory depression, which related to Brain Derived Neurotrophic Factor (BDNF). Even though level of peripheral BDNF is closely related to depression treatment, the investigators still have little idea on role of BDNF. In this research, the investigators are going to find the genetic variation affecting treatment response and process, figure out specific role of BDNF in depressive patient correlated with Neuroimaging. Along with BDNF, many kinds of proinflammatory cytokine showed increased amount related to depressive patient. Leptin, adiponectin, and plasma tryptohphan are also seen to be related to response of depression. Here, the investigators are trying to see specific difference on neuroimaging shown in depressive patient related to peripheral marker. The investigators will evaluate the 36 depressive patients compared to 24 normal control. For depressive patients, after excluding other bipolar spectrum disorder, psychotic disorder, other neurocognitive disorder, subjects who have organic brain lesion, tested as HAM D score above 16, will be included in this research. As a psychiatric evaluation, the investigators will do the MINI International Psychiatric Interview Plus (MINI Plus), Suicidal ideation evaluation, Hamilton Depression Inventory 17 (HAM D 17), Hamilton Anxiety Inventory (HAM A) to get the information of their clinical severity. As a neuroimaging evaluation, the investigators will do the magnetic resonance imaging (MRI) with diffusion tensor imaging and amyloid Positron Emission Tomography(PET) to see the specific deposition. For peripheral marker for inflammation and other neurotrophic factor, the investigators will do the platelet BDNF level,and other pre-inflammatory factors. The investigators will also check for genotyping for BDNF. For follow up evaluation, the investigators will keep up the psychiatric evaluation with HAM D, HAM A and peripheral proteinomic evaluation with platelet BDNF level, and other pro-inflammatory cytokines.

This research will figure out the correlation between neurotrophic factor as BDNF, and inflammatory factor seen in peripheral blood assay with treatment response in depression. Also the investigators are trying to integrate the peripheral change along with BDNF genotyping and specific change seen in neuroimaging. Replicating this research with high statistical power would be promising to find 'reliable peripheral marker for prognosis of depression'.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as major depressive disorder with MINI and DSM-5 criteria whose age is more than 65 years
* Whose score of Hamilton Depression Scale is more than 16
* Whose first depressive episode onset was later than one's age of 60
* Who is free from antidepressants for 2 weeks

Exclusion Criteria:

* Subjects with past history of Psychotic disorder or with present symptoms related to psychotic disorders
* Bipolar Spectrum Disorder
* With Neurocognitive disorder such as Parkinson's disease, Huntington's chorea, Mild Cognitive Disorder, or Dementia
* Who ever diagnosed as a Cognitive disability
* Who have serious medical condition which needs to be cared (e.g, cancer)
* Who have past history of epileptic disorder or present with epileptic disorder in treatment
* Who have recent history of alcohol or other substance use disorder within 6 months and suspicious for this condition
* Who is suspicious for the clinically implicable personality disorder
* Who is suspicious for the brain injury
* Who is having trouble with uncontrolled claustrophobia, hard to go through neuroimaging

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older than 65 years free from other main psychiatric diagnosis except major depressive disorder free from neurocognitive disorder
  normal control: older than 65 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The change of Psychiatric symptom profile scores | baseline, 1month, 3months
  Hamilton depression inventory 17 (HAM-D), Hamilton anxiety inventory (HAM-A) and peripheral proteinomic evaluation

SECONDARY OUTCOMES:
The change of subjective Cognitive decline assessment profiles | baseline, 1month follow up, 3 months follow up, cognitive function assessment with subjective one and objective one

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jin Jeon, M.D.,Ph.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No